CLINICAL TRIAL: NCT01565525
Title: Can Changing How Moms Eat Prevent Obesity in Toddlers?
Brief Title: Anticipatory Guidance to Prevent Childhood Obesity
Acronym: MOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Judith Groner, Clinical Professor of Pediatrics, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HD50944
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Childhood Obesity
Keywords: well child visit; anticipatory guidance; obesity prevention; infant feeding
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bright Futures (No Intervention): This represents 'usual care' in the pediatric office. The anticipatory guidance regarding nutrition is based on the Bright Futures Pocket Guide.
- Maternal focused intervention (Experimental): Childhood obesity prevention was approached in this arm via anticipatory guidance aimed at maternal eating habits.
  Interventions: Behavioral: Maternal focused intervention
- Ounce of Prevention (Active Comparator): This is a program of anticipatory guidance given to mothers of infants ages 2 weeks to one year which focuses on serving size per age and tips for introducing new foods for the infant.
  Interventions: Behavioral: Ounce of Prevention

INTERVENTIONS:
Behavioral: Maternal focused intervention — This is a series of information given to mothers at child's well child visits (6 in all) starting at the newborn visit focused in maternal eating habits, using the mother as a potential 'agent of change' for the family and infant in modeling healthy eating habits.
  Other Names: MOMS
  Arms: Maternal focused intervention
Behavioral: Ounce of Prevention — This intervention is given via a series of handouts given to mothers at their child's well visit from newborn period to one year of age, focusing on serving size and frequency and the introduction of new foods.
  Other Names: "Ounce"
  Arms: Ounce of Prevention

SUMMARY:
The purpose of this pilot project is to test anticipatory guidance, which is information given to families during a well child visit to prevent obesity during childhood. The objectives were to compare two styles of anticipatory guidance during the first year of life, maternal focused and infant focused, versus usual care and determine which style, if any, showed the most ideal infant feeding behaviors at age 1 year and to see if there were any differences in infant weight for height at one year of age. The investigators hypothesized that mothers who received the maternal focused anticipatory guidance (which gave information on eating family meals, not having tv on during meals, and maternal nutrition) would actually have the best infant feeding behaviors and weight for height of infants at one year.

ELIGIBILITY:
Inclusion Criteria:

Maternal/infant pairs Infant under 2 months of age Mother English speaking

Exclusion Criteria:

History of Neonatal ICU stay in infant Gestation less than 37 weeks in infant chronic disease in infant known genetic disorder in infant foster care placement in infant

Ages: 2 Weeks to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2005-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Infant weight for height | One year after study entry
  Infant weight for height will be assessed to see if proportions of elevated weight for height are lower in intervention groups as compared to usual care.

SECONDARY OUTCOMES:
Maternal feeding behaviors | One year after study entry.
  Several maternal feeding behaviors, including amount of vegetables and fruit offered to infant, eating as a 'family', amount of television watching by the infant, and juice intake by the infant were secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Groner, MD, Principal Investigator — Nationwide Children's Hospital, Columbus Ohio
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Groner JA, Skybo T, Murray-Johnson L, Schwirian P, Eneli I, Sternstein A, Klein E, French G. Anticipatory guidance for prevention of childhood obesity: design of the MOMS project. Clin Pediatr (Phila). 2009 Jun;48(5):483-92. doi: 10.1177/0009922809331799. Epub 2009 Feb 25. PMID 19246415
- [Background] Nicholson LM, Schwirian PM, Klein EG, Skybo T, Murray-Johnson L, Eneli I, Boettner B, French GM, Groner JA. Recruitment and retention strategies in longitudinal clinical studies with low-income populations. Contemp Clin Trials. 2011 May;32(3):353-62. doi: 10.1016/j.cct.2011.01.007. Epub 2011 Jan 27. PMID 21276876
- [Derived] French GM, Nicholson L, Skybo T, Klein EG, Schwirian PM, Murray-Johnson L, Sternstein A, Eneli I, Boettner B, Groner JA. An evaluation of mother-centered anticipatory guidance to reduce obesogenic infant feeding behaviors. Pediatrics. 2012 Sep;130(3):e507-17. doi: 10.1542/peds.2011-3027. Epub 2012 Aug 13. PMID 22891225